CLINICAL TRIAL: NCT02102971
Title: Autophagy in Liver Injury: Changes in Autophagy Biomarkers During Liver Surgery
Brief Title: Observational Study of Biomarker During Liver Surgery
Status: Terminated | Type: Observational
Why Stopped: Expired with UF IRB.
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400182 -N; R01DK079879 (NIH)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Liver Cancer; Hepatobiliary Tract Adenomas and Carcinomas
Keywords: liver; ischemia; reperfusion
MeSH Terms: conditions — Liver Neoplasms; Carcinoma; Ischemia | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — liver tissues during liver surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatocellular carcinoma: Participants undergoing a liver resection/liver transplantation surgery. During the liver surgery a small piece of tissue will be removed to undergo additional laboratory testing.
  Interventions: Procedure: Hepatocellular carcinoma

INTERVENTIONS:
Procedure: Hepatocellular carcinoma — Participants undergoing a liver resection/liver transplantation surgery. During the liver surgery a small piece of tissue will be removed to undergo additional laboratory testing.
  Other Names: Liver resection; Liver transplantation surgery

SUMMARY:
The investigators would like to study whether Sirtuin 1 (SIRT1) plays a cytoprotective role in liver ischemia/reperfusion, and ultimately to develop therapeutic strategies to improve hepatic function of patients with liver diseases.

DETAILED DESCRIPTION:
If asked to participate in this research study, it is because a liver resection/liver transplantation surgery has been scheduled. During the procedure a small section will be collected for additional testing of Sirtuin 1. In addition, information concerning the liver disease, laboratory and pathology results after surgery will be collected by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* liver resection > 2 segments,
* plate count > 100 x 109/L, and
* prothrombin activity >60%.

Exclusion Criteria:

* liver cirrhosis,
* portal hypertension,
* steatohepatitis or severe steatosis,
* patients receiving additional ablation therapies,
* laparoscopic resection, and
* simultaneous extrahepatic procedures such as colorectal resection or pancreatoduodenectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver Disease Requring Liver Resection Surgery
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-10; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Biochemical analysis of sirtuin1 from liver tissues during liver surgery | 30 minutes during liver surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Sung Kim, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No